CLINICAL TRIAL: NCT01984190
Title: ActiveCare+S.F.T® Outcomes Registry (ACOR)
Brief Title: Multicenter Registry for Effectiveness Analysis of ActiveCare+S.F.T® Mobile Compression Device for Thrombosis Prevention in Hip and Knee Arthroplasty
Acronym: ACOR
Status: Completed | Type: Observational
Sponsor: Medical Compression Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: Version date: 9 -8 -10
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2013-11

CONDITIONS: Venous Thromboembolism
Keywords: venous thromboembolism; deep vein thrombosis; pulmonary emboli; hip arthroplasty; knee arthroplasty; efficacy; mobile compression device; mechanical device; prophylaxis.
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lower Extremity Joint Arthroplasty: Postoperative venous thromboembolism incidence in lower extremity joint arthroplasty using only the mobile compression device with or without aspirin for venous thromboembolism prevention. Sub-analysis of Total Hip Arthroplasty and Total Knee Arthroplasty will be included.

SUMMARY:
Venous thromboembolic events (VTE), either deep vein thromboses or pulmonary emboli, are important complications in patients undergoing knee or hip arthroplasty. This multicenter Clinical Registry is aimed at collecting large volume clinical effectiveness data of ActiveCare+S.F.T® mobile compression device +/- aspirin in lowering the potential risk of venous thromboembolism (VTE) prophylaxis in patients undergoing primary lower extremity total joint arthroplasty. The results can then be compared to pharmacology protocols.

DETAILED DESCRIPTION:
Orthopaedic surgeons at ten sites in the United States will participate in a registry to collect postoperative venous thromboembolism incidence in lower extremity joint arthroplasty patients using the mobile compression device. Patients will be included in the registry if they are eighteen years of age or older and undergoing primary unilateral hip arthroplasty (including hip resurfacing) or primary unilateral knee arthroplasty (including unicondylar knee arthroplasty) using only the mobile compression device with or without aspirin for venous thromboembolism prevention. Patients will be excluded if they are scheduled for a revision surgery, have a history of venous thromboembolism, a coagulation disorder, a solid tumor malignancy within the last five years, or had a major surgery in the three months prior to the joint surgery. An attempt to enroll every patient consecutively will be made at each institution and only those patients who did not meet the inclusion criteria or declined participation will not be included. Use of the ActiveCare+S.F.T® mobile compression device will begin intra-operatively and continue for a minimum of 10 days. The decision to use aspirin is at the discretion of each surgeon. All patients will be evaluated within three months postoperatively, documenting evidence of deep venous thrombosis or pulmonary emboli.

1. Registry Procedures

   * Patients will complete a 1 page questionnaire regarding their usage of the mechanical compression device. The de-identified information from the questionnaire will be entered into a web based computer database by a research coordinator at each of the ten sites. The web based registry was created by a third party (Global Visions Technology, Inc.).
   * Once the study is closed to enrollment and data entry is complete, the database manager will pull all the data from the web based registry and import into a statistical software program for analysis.
   * A power analysis found that sample sizes of 1500 in the device group and any drug group would be sufficient to achieve power in excess of 90% to detect a non-inferiority margin difference between the venous thromboembolism proportions in the two groups of 1.0%. In these calculations, we considered drug group venous thromboembolism rates between 0.5% and 1.0% and the device group venous thromboembolism rate was taken to be the drug group rate +1.0% under the null hypothesis of inferiority. Power was computed for the case when the actual device venous thromboembolism rate was identical to the drug comparator rate. The test statistic used was the one-sided score test, with the significance level set at 0.025.
   * SPSS version 13.0 (SPSS, Chicago, Illinois) and NCSS Version 7.1.21 (NCSS LLC, Kaysville, Utah) will be used for analysis of the registry data. Means will be calculated to describe continuous variables (age, height, weight) and frequencies will be calculated to describe categorical variables (surgery type, aspirin use, incidence of symptomatic venous thromboembolism). Upper bound 97.5% CIs will be calculated around the observed venous thromboembolism rate difference between the mobile compression device and each drug comparator.
2. Quality Factors

   * Institutional Review Board (IRB)approval will be obtained at each site.
   * Patient privacy will be protected per the Health Insurance Portability and Accountability Act (HIPAA). Patients will remain anonymous; all patient identifiers will be purged from the data at the originating center. Patient care will NOT be affected in any way by participation in the study.
   * Accounts were set up for each coordinator with respective passwords for security. A data entry guide will be distributed to each coordinator, which will give instructions for entering each variable. Additionally, each coordinator will be required to view an instructional video online before they will be permitted to begin data entry into the registry.
   * Validation criteria will be set up for each field so that data are entered in the correct format (eg, must enter four digits for the year, sex must be entered as "M" or "F", etc). Ranges will be constructed to minimize data entry errors (eg, "number of days the device was worn" will be restricted to a number between 0 and 15 only). If any required fields are left blank, a prompt will come up to ask the coordinator to fill in the missing data. The record will be marked as incomplete until all required fields are completed. Each of the 10 sites will only have access to view their own data.
   * Periodic data checks will be performed by the database manager, who will query all fields and to keep track of how enrollment is going at each site. When the study is closed, the database will be locked by the database manager.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (Age >18 yrs).
* Patient intended to undergo elective primary unilateral total hip arthroplasty (THA) or total knee arthroplasty (TKA), or unicondylar knee arthroplasty (UKA).
* Patient is using only ActiveCare+S.F.T® +/- aspirin for venous thromboembolism (VTE) prevention(Aspirin (ASA) can be prescribed at the discretion of the surgeon).

Exclusion Criteria:

* Patient with known coagulation disorder
* Patient currently treated with anticoagulant medications.
* Patients with current signs and symptoms of or history of deep vein thrombosis(DVT) or pulmonary embolism (PE).
* Patients currently suffering from a solid tumor malignancy.
* Patients who underwent major surgery procedure within 3 months prior to participation in the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will include all Adult patients scheduled for elective unilateral total hip arthroplasty (THA) or total knee arthroplasty (TKA), or unicondylar knee arthroplasty (UKA), where the orthopaedic surgeon is using the ActiveCare+S.F.T® mobile compression device as a monotherapy for venous thromboembolism prevention.
Sampling Method: Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Incidence of deep venous thrombosis or pulmonary emboli | Within 3 months post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Clifford W Colwell, Jr., MD, Principal Investigator — Shiley Center for Orthopaedic Research and Education at Scripps Clinic
Locations (10):
- United States (10):
  - Arkansas Specialty Orthopaedics, Little Rock, Alaska
  - Shiley Center for Orthopaedic Research and Education at Scripps Clinic, La Jolla, California
  - VA Palo Alto Health Care System, Menlo Park, California
  - Rubin Institute for Advanced Orthopedics,, Baltimore, Maryland
  - Twin Cities Orthopaedics, Edina, Minnesota
  - Washington University School of Medicine, Department of Orthopaedic Surgery, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The Center Orthopedic & Neurosurgical Care &Research, Bend, Oregon
  - Anderson Orthopaedic Clinic, Alexandria, Virginia

REFERENCES:
- [Background] Colwell CW Jr, Froimson MI, Mont MA, Ritter MA, Trousdale RT, Buehler KC, Spitzer A, Donaldson TK, Padgett DE. Thrombosis prevention after total hip arthroplasty: a prospective, randomized trial comparing a mobile compression device with low-molecular-weight heparin. J Bone Joint Surg Am. 2010 Mar;92(3):527-35. doi: 10.2106/JBJS.I.00047. PMID 20194309
- [Result] Colwell CW Jr, Froimson MI, Anseth SD, Giori NJ, Hamilton WG, Barrack RL, Buehler KC, Mont MA, Padgett DE, Pulido PA, Barnes CL. A mobile compression device for thrombosis prevention in hip and knee arthroplasty. J Bone Joint Surg Am. 2014 Feb 5;96(3):177-83. doi: 10.2106/JBJS.L.01031. PMID 24500578